CLINICAL TRIAL: NCT06135740
Title: Impact of Notifications on Nutrition, Sleep, and Physical Activity on Intellectual Function and Muscle Mass in OldeR Adults (INSPIOR)
Brief Title: Impact of Nutrition, Sleep, and Physical Activity on Intellectual Function and Muscle Mass in Older Adults
Acronym: INSPIOR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Tokyo University (Other)
Collaborators: Google LLC. (Industry)
Responsible Party: Principal Investigator, Tatsuhiro Hisatsune, Associate Professor, Tokyo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 22-360
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Cognition Disorders in Old Age; Cognitive Function; Frailty/Sarcopenia; MCI
MeSH Terms: conditions — Frailty; Sarcopenia

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Notification on Nutrition, Sleep, and Physical Activity based on fitbit-based data
  Interventions: Device: Fitbit wearing, with notification for sleep, activity and nutrition based fitbit data
- Control (Sham Comparator): Regular Care
  Interventions: Device: Routine care

INTERVENTIONS:
Device: Fitbit wearing, with notification for sleep, activity and nutrition based fitbit data — Notification on Nutrition, Sleep, and Physical Activity based on fitbit-based data, and Nutritional supplementation and Promotion of Exercise
  Arms: Intervention
Device: Routine care — Regular Care on sleep, activity and nutrition
  Arms: Control

SUMMARY:
The goal of this prospective, single site, interventional randomized control trial is to treat age related health conditions in adults older than 65 years and functional independence. The main question of the study is to answer the effectiveness of notification on activity, sleep, and nutrition based on wearable device Fitbit recorded data for the improvement of health conditions including intellectual property and physical function, compared to usual care. Participants in the intervention arm will be given a Fitbit Charge 5 device and asked to wear this for the duration of the study, including during sleep. The study intervention will run for 6 months. Notifications will be issued using a monitoring software in Japanese, and issued automatically to participants. Participants in the control arm will be given a routine care and health-related information. Researchers will compare cognitive performance, muscle mass and physical activity between the two groups to see if the notification based on Fitbit data would promote the health conditions of older adults.

DETAILED DESCRIPTION:
This is a prospective, single site, interventional randomized control trial. The primary purpose is to treat age related health conditions. The current study is nested within an established cohort based in Kashiwa City in Japan, which consists of older adults living independently. The inclusion criteria of this study is age equal to or older than 65 years and functional independence (i.e., not requiring nursing care provided by long-term care insurance). The investigators plan to conduct a randomized controlled trial to test the effectiveness of notification based on Fitbit recorded data, used to prompt health and wellness actions on a variety of health outcomes, compared to usual care. On enrollment, baseline demographic and health information as well as baseline measurements for quality of life, and physical and mental health, will be collected. Subsequently, the study intervention will run for 6 months. Participants in the intervention arm will be given a Fitbit Charge 5 device and asked to wear this for the duration of the study, including during sleep. Participants will receive sessions to teach them how to use the Charge 5 device and access the information produced. Those who meet the above criteria for intervention will receive automatically generated notifications that include lifestyle recommendations. Notifications will be issued using a monitoring software in Japanese, and issued automatically as text alerts to participants. Participants will receive encouraging notifications to promote adherence and health condition. Participants in the control arm will be given a routine care and health-related information. Participants who fail to exhibit a behavior change in the week following the alert, or who are not engaging with the study (e.g., by not wearing the Fitbit device) will be followed up by phone by a member of the community research group. Researchers will compare cognitive performance and physical activity between the two groups to see if the notification based on Fitbit data would promote the health conditions of older adults. Results of this trial will be valuable for informing further implementation of wearable devices and related digital devices in elderly populations in Japan and other countries in the region.

ELIGIBILITY:
Inclusion Criteria:

* Over 65 years of age.
* Living in Japan.
* Living independently with or without carer support.
* Able and willing to wear a Fitbit for the duration of the study (≥20 hours a day, including during sleep).
* Individuals that are able and willing to receive and act on interventions.
* Has capacity to consent to inclusion in the study.
* Smartphone access to allow Fitbit installation and setup.
* Has one or more of the following comorbidities:

  * BMI <20 (65-69 years), <21.5 (≥70 years)
  * Pre-frail or Frail: scoring 1-2 (pre-frail) or 3+ (frail) based on the FRAIL questionnaire
  * Sarcopenia: low grip strength (female <18 kg, male <28 kg); Gait speed (< 1m/s); low Skeletal Muscle mass Index (female 5.7 kg/m2; male 7 kg/m2)

Exclusion Criteria:

* Individuals receiving full time care in a care facility.
* Individuals that are unable to receive and/or act on interventions.
* Individuals who are existing wearable users, or who have prior experience using a wearable to manage their health.
* Individuals with uncontrolled hypertension, diabetes, CKD or with cardiac pacemakers and/or cardiovascular stent(s).
* Individuals who have any additional condition or situation that the Investigator (PI) or designee determines as inappropriate for participation in this study.
* Individuals with no comorbidities as defined above.

Ages: 65 Years to 92 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2023-11-08 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Executive function | 0 - 6 months
  TMT
General Cognition | 0 - 6 months
  MoCA
Muscle mass | 0 - 6 months
  Skeletal Muscle mass Index

SECONDARY OUTCOMES:
Amount of exercise | 0 - 6 months
  Step counts measured by fitbit
Amount of sleep | 0 - 6 months
  Total sleep time measured by fitbit

OTHER OUTCOMES:
Frail/Sarcopenia | 0 - 6 months
  Frailty index
Malnutrition | 0 - 6 months
  Protein intake

CONTACTS AND LOCATIONS:
Overall Officials: Tatsuhiro Hisatsune, PhD, Principal Investigator — Associate Professor
Locations (1):
- Graduate School of Frontier Sciences, The University of Tokyo, Kashiwa, Chiba, Japan